CLINICAL TRIAL: NCT06966804
Title: Efficacy of Alpha Blockers (Terazosin vs Tamsulosin) in Reducing Ureteral Stent Related Symptoms - An Open-label, Randomized Controlled Trial
Brief Title: Comparison of Alpha Blockers (Terazosin and Tamsulosin) in Reducing Ureteral Stent Related Symptoms
Acronym: TRAM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Penang Hospital, Malaysia (Other Government)
Responsible Party: Principal Investigator, Ooi Yeon Wee, Doctor, Penang Hospital, Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRR-24-03594-URB; RSCH ID-24-05599-H07 (Other: National Medical Research Registry)
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Stent Related Symptoms
Keywords: alpha blockers; ureteral stent-related symptoms; tamsulosin; terazosin; USSQ
MeSH Terms: interventions — Terazosin; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Terazosin (Experimental): Terazosin 2mg ON
  Interventions: Drug: Terazosin
- Tamsulosin (Experimental): Tamsulosin 0.4mg ON
  Interventions: Drug: Tamsulosin
- Standard care (No Intervention): No medication

INTERVENTIONS:
Drug: Terazosin — Subject will complete 14-day course of Terazosin
  Arms: Terazosin
Drug: Tamsulosin — Subject will complete 14-day course of Tamsulosin
  Arms: Tamsulosin

SUMMARY:
The goal of this clinical trial is to compare how well Terazosin, Tamsulosin and standard care (no alpha-blocker) reduce urinary symptoms after ureteral stent placement. This trial also learn about the safety of these two study medications.

Main objective:

• To compare how well Terazosin, Tamsulosin and standard of care reduce post-stenting urinary symptoms.

Secondary objectives:

* To compare painkiller use among the groups.
* To assess differences in Body pain, General health, Work performance, Sexual matters, and Additional problems using a questionnaire (USSQ).
* To assess differences in side effects.

After stent placement, subjects will be randomly assigned to one of three groups:

1. Terazosin (alpha-blocker) for 14 days
2. Tamsulosin (alpha-blocker) for 14 days
3. Standard of care (no alpha-blocker). All subjects will be discharged with standard pain-killers and a diary to track usage. Subjects in Terazosin and Tamsulosin groups will receive respective study medications to complete 14 days course of treatment.

Follow-Up:

* Day 7: A phone call will check medication use and any side effects.
* Day 15: Clinic visit for stent removal (standard practice). Subjects will complete the USSQ questionnaire, and medication compliance will be reviewed.

End of study: Final phone call to check for any additional side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Malaysian age 18 years old and above.
2. Able to provide written informed consent to participate in the trial.
3. Willing to comply with study procedures.
4. Unilateral intracorporeal lithotripsy procedure with ureteral stent placement for uncomplicated ureteric or renal calculi

Exclusion Criteria:

1. Known comorbidity that increase the risk of complication

   1. Prostate pathology: Benign prostate hyperplasia, prostatitis, prostatic carcinoma
   2. Bladder pathology: Bladder tumor, stone, overactive bladder
   3. Ureteral abnormality/ trauma, urethral stricture
   4. Concomitant urinary tract infection
   5. Orthostatic hypotension
   6. Solitary kidney
2. Previous pelvic/ gynaecological surgery
3. Patient is concomitantly receiving treatment from a pain clinic for chronic pain management.
4. Pregnancy (for women of childbearing potential)
5. Known history of allergic reactions to tamsulosin or terazosin
6. Patient is concomitantly taking warfarin or H2 receptor blockers
7. Patients with clinical condition(s) judged by the researcher/ clinician to be unsuitable for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
To determine the efficacy of Terazosin, Tamsulosin and standard of care in reducing post-stenting urinary symptoms | From randomization to the end of the treatment at 14 days
  Ureteral Stent Symptom Questionnaire (USSQ)- "Urinary Symptom score" domain. This domain focuses on issues related to urine storage and voiding, including symptoms such as weak stream, intermittent, incomplete empty, straining to start, frequency of spasm, urgency, nocturia, dysuria, hematuria, urge incontinence and impact quality of life.
  Each symptom is scored, with higher score indicating more severe symptoms. The total score ranges from 11 ( best outcome) to 56 (worst outcome).

SECONDARY OUTCOMES:
To determine the difference in analgesic requirement | From randomization to the end of the treatment at 14 days
  Analgesic usage from patient's analgesic diary. Patients will be discharged with a standardized institutional analgesic regimen. Daily analgesic use will be recorded in a patient diary, and total consumption will be calculated at the end of the treatment period.
  The total analgesic dose will be compared across the three study arms. A higher total analgesic requirement will indicate more severe stent-related symptoms.
To determine the efficacy of Terazosin, Tamsulosin and standard of care in reducing post-stenting: Body pain, General health Work performance, Sexual matters, Additional problems | From randomization to the end of the treatment at 14 days
  Ureteral Stent Symptom Questionnaire (USSQ) Domains
  Higher scores indicate worse outcomes across all domains:
  1. Body Pain Score: Assesses pain in loin/flank, hypochondrium, groin, bladder, external genitalia, and kidney area during voiding/activity.
  2. General Health: Evaluates physical symptoms, vitality, psychosocial impact, dependence on others, social life enjoyment, and activity limitations.
  3. Work Performance: Measures absenteeism, productivity loss, concentration issues, functional limitations and overall work quality.
  4. Sexual Matters: Assesses pain during intercourse, satisfaction, and complete sexual dysfunction.
  5. Additional Problems: Identifies post-insertion complications.
  6. Global Quality of life with stent in situ: Determines willingness for future stenting, reflecting overall tolerance.
To describe the difference in adverse events | From randomization to the end of the treatment at 14 days
  Collect adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- Malaysia (2):
  - Sultanah Bahiyah Hospital, Alor Setar, Alor Star, Kedah
  - Hospital Pulau Pinang, George Town, Pulau Pinang